CLINICAL TRIAL: NCT03551210
Title: An International, Multicenter, Randomized, Double-blind, Double-dummy, Two-way, Parallel Group, Controlled Study to Compare the Efficacy and Safety of Intravenous and Oral Nemonoxacin Versus Tavanic® in Adult Patients With Community-acquired Pneumonia
Brief Title: Efficacy and Safety of Nemonoxacin vs Levofloxacin in Adult Patients With Community-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: OCT Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CJ01060044
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Pneumonia, Bacterial
Keywords: nemonoxacin; community-acquired pneumonia; quinolones
MeSH Terms: conditions — Pneumonia, Bacterial; Community-Acquired Pneumonia | interventions — nemonoxacin; Ofloxacin; Levofloxacin

STUDY DESIGN:
Intervention Model Description: All eligible patients will be randomized to receive either treatment with Nemonoxacin or Tavanic® in a ratio of 1:1.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nemonoxacin (Experimental): Nemonoxacin solution for infusion, 500 mg (250 ml), daily, as single intravenous infusion over 90-110 minutes followed by infusion of Placebo (100 ml), solution for infusion, over a minimum duration of 60 minutes.
  Then will be switched to oral therapy with Nemonoxacin capsules, 500 mg once daily (two 250 mg capsules).
  Interventions: Drug: Nemonoxacin; Drug: Placebo (100 ml)
- Tavanic® (Active Comparator): Tavanic® solution for infusion, 500 mg (100 ml), daily, as single intravenous infusion over a minimum duration of 60 minutes with previous infusion of Placebo (250 ml), solution for infusion, over 90-110 minutes.
  Then will be switched to oral therapy with Tavanic®, over-encapsulated film coated tablets, 500 mg once daily (two capsules each containing 250 mg film coated tablet).
  Interventions: Drug: Tavanic; Drug: Placebo (250 ml)

INTERVENTIONS:
Drug: Nemonoxacin — Solution for infusion, 500 mg (250 ml)
  Arms: Nemonoxacin
Drug: Nemonoxacin — Capsules, 250 mg
  Arms: Nemonoxacin
Drug: Tavanic — Solution for infusion, 500 mg (100 ml)
  Other Names: Levofloxacin
  Arms: Tavanic®
Drug: Tavanic — Film coated tablets (each tablet is placed into a capsule shell (overencapsulated) for blinding purposes), 250 mg
  Other Names: Levofloxacin
  Arms: Tavanic®
Drug: Placebo (250 ml) — 0.9% NaCl (250 ml), solution for infusion
  Arms: Tavanic®
Drug: Placebo (100 ml) — 0.9% NaCl (100 ml), solution for infusion
  Arms: Nemonoxacin

SUMMARY:
The primary objective of this study was to evaluate the clinical efficacy of treatment with Nemonoxacin compared with Tavanic® in patients with community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
Treatment-naive patients with CAP and patients with treatment failure were screened and if met the eligible criteria were randomized to receive either treatment with investigational product or comparator. Patients started to receive intravenous therapy with Nemonoxacin or Tavanic® and then upon a decision of investigator patients were switched to oral therapy with the same product.

Intravenous therapy included two consequence infusions (antibiotic solution and placebo solution) to maintain blinding. Intravenous therapy should have been given for at least 3 days and could have been prolonged by a decision of investigator up to 7 days. Then investigator switched a patient from intravenous to oral therapy on Day 4(8) of the study if the specific criteria of clinical stability were achieved. To maintain blinding during oral antibiotic therapy each Tavanic® tablet was placed into a capsule shell (over-encapsulated), that was identical in appearance to a Nemonoxacin-containing capsules.

The average duration of treatment (including intravenous and oral therapy) for each patient was 7(14) days and during this period patients should have stayed at hospital. After completion of the treatment patients could have been discharged from the hospital and returned for examinations within 1-2 days after the last dose (end of treatment visit). Then the patients attended the investigational site within 7-9 days after the last dose (test of cure visit). Then the investigator contacted the patients by phone within 21-23 days after the last dose (long-term follow-up visit).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient.
* Patients with moderate to severe community-acquired pneumonia who need inpatient treatment but do not need intensive care unit treatment.
* The presence of at least 3 of the following symptoms / signs:

  1. cough;
  2. purulent sputum production;
  3. tachypnea (respiratory rate > 24 breathes/minute);
  4. chills;
  5. fever (rectal / tympanic temperature ≥ 38.5°C or axillary / oral / skin temperature ≥ 38.5°C);
  6. white blood cells (WBC) count of ≥ 10.0 x 10^9/L or ≥ 15% immature neutrophils (bands; regardless of peripheral WBC count).
* Radiological evidence of (a) new infiltrate(s) consistent with bacterial pneumonia at baseline.
* Treatment-naive patients or patients who have received single dose of a short-acting antibacterial drug within 24 hours of enrollment or patients with treatment failure who have received antibiotics (with the exception of quinolones or fluoroquinolones) for less than 72 hours.
* Consent to use contraception during participation in the study (for women of childbearing potential and men).

Exclusion Criteria:

* Known hypersensitivity to quinolones, fluoroquinolones or any of the excipients.
* Female patients who are pregnant or nursing.
* History of tendon disease / disorder related to quinolone treatment.
* Known congenital or documented-acquired QT / QTc(F) prolongation on ECG (QTc(F) interval more than 450 ms); concomitant use of drugs, reported to increase the QT interval; uncorrected hypokalaemia and uncorrected hypomagnesemia; clinically relevant bradycardia; clinically relevant heart failure with reduced left-ventricular ejection fraction; previous history of symptomatic arrhythmias.
* History of bronchiectasis, cystic fibrosis, bronchial obstructions excluding chronic obstructive pulmonary disease.
* History of epilepsy and/or history of psychotic disorder.
* Patients with history of myasthenia gravis.
* Patients with diabetes mellitus.
* Known glucose-6-phosphate dehydrogenase deficiency.
* Active hepatitis or decompensated cirrhosis.
* Alanine transaminase or aspartate transaminase increase > 3 fold upper limit of normal (ULN).
* Patients with creatinine ≥ 1.1 fold ULN.
* Patients requiring concomitant systemic or inhaled antibiotics (e.g., tobramycin).
* Known or suspected active tuberculosis or endemic fungal infection.
* Concomitant immunosuppressive therapy including a long-term (more than 2 weeks) treatment with oral or intravenous glucocorticoids at doses of 20 mg and higher of prednisone daily or an equivalent dose of other glucocorticoids.
* Patients known to have HIV-positive status or AIDS or known to have other disease that seriously affects the immune system such as active haematological or solid organ malignancy, or splenectomy.
* History of drug or alcohol abuse.
* Patients have received quinolones or fluoroquinolones within 14 days before enrollment.
* Previous enrolment in this study or participation in another study within the previous 4 weeks.
* Patients with any severe medical condition as determined by medical history that, in the opinion of the investigator, does not allow the patient to carry out all planned procedure of the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (25):
- Russia (25):
  - Regional budget healthcare institution "Ivanovo regional clinical hospital", Ivanovo
  - City clinical hospital #1 n.a. N.I. Pirogov of Moscow Healthcare Department, Moscow
  - City Clinical hospital n.a. V. V. Vinogradov, Moscow
  - FSOE Main Military Clinical Hospital n.a. academician N.N. Burdenko of the Ministry of Defence of the Russian Federation, Moscow
  - SBHI Moscow City clinical hospital # 15 n.a. O.M. Filatov of Moscow Healthcare Department, Moscow
  - City Clinical Hospital #25, Novosibirsk
  - City clinical hospital #2, Novosibirsk
  - SBHI of Novosibirsk region City Clinical Hospital of Emergency Medical Care №2, Novosibirsk
  - Republic Hospital named after V.A. Baranov, Petrozavodsk
  - Pskov regional clinical hospital, Pskov
  - Baltic Medicine LLC, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - City hospital #38 n.a. N.A. Semashko, Saint Petersburg
  - Mariinsky City Hospital, Saint Petersburg
  - Multidisciplinary City Hospital # 2, Saint Petersburg
  - Scientific Research Institute of Influenza of the Ministry of Healthcare of Russian Federation, Saint Petersburg
  - Regional clinical hospital, Saratov
  - Clinical hospital of emergency medical care, Smolensk
  - Scientific Research Institute of Antimicrobial Therapy of Smolensk State Medical University, Smolensk
  - Siberian State Medical University of the Ministry of Healthcare of Russian Federation, Tomsk
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Voronezh Regional Clinical Hospital #1, Voronezh
  - Central city hospital #7, Yekaterinburg
  - City clinical hospital #40, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of subjects was conducted by 25 clinical sites in Russia between May 2016 and 2017. Totally 356 patients were screened and 342 eligible patients were randomized to receive Nemonoxacin or Tavanic in 1:1 ratio (171 subjects in each group).
Groups:
- Nemonoxacin: Nemonoxacin solution for infusion, 500 mg (250 ml), daily, as single intravenous infusion over 90-110 minutes followed by infusion of Placebo (100 ml), solution for infusion, over a minimum duration of 60 minutes.
  Then will be switched to oral therapy with Nemonoxacin capsules, 500 mg once daily (two 250 mg capsules).
  Nemonoxacin: Solution for infusion, 500 mg (250 ml)
  Nemonoxacin: Capsules, 250 mg
  Placebo (100 ml): 0.9% NaCl (100 ml), solution for infusion
- Tavanic®: Tavanic® solution for infusion, 500 mg (100 ml), daily, as single intravenous infusion over a minimum duration of 60 minutes with previous infusion of Placebo (250 ml), solution for infusion, over 90-110 minutes.
  Then will be switched to oral therapy with Tavanic®, over-encapsulated film coated tablets, 500 mg once daily (two capsules each containing 250 mg film coated tablet).
  Tavanic: Solution for infusion, 500 mg (100 ml)
  Tavanic: Film coated tablets (each tablet is placed into a capsule shell (overencapsulated) for blinding purposes), 250 mg
  Placebo (250 ml): 0.9% NaCl (250 ml), solution for infusion
Period: Overall Study
Arm/Group | Nemonoxacin | Tavanic®
Started | 171 | 171
Completed | 161 | 151
Not Completed | 10 | 20
Not completed — Adverse Event | 5 | 6
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Needed in other antibiotic treatment | 2 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Absence of visit 4 and 5 | 1 | 0
Not completed — No drug for dispensing | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-To-Treat population (mITT) - all randomized patients received at least one dose of investigational drugs, in compliance with at lest minimal disease criteria (inclusion criteria 3 and 4) and had at least one assessment of clinical efficacy in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Nemonoxacin | Tavanic® | Total
Number analyzed (Participants) | 169 | 166 | 335
Age, Continuous [Mean (Full Range); unit: years] | 42.0 [18 to 69] | 43.3 [18 to 70] | 42.6 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 132
  Male | 103 | 100 | 203
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  European | 168 | 166 | 334
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Calculated as patient's weight (kg)/height (m^2)
  kg/m^2 | 25.4 (5.4) | 26.1 (5.6) | 25.8 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Success as Judged by the Investigator
Description: Clinical response is evaluated as clinical success if: all signs and symptoms of pneumonia are resolved or improved with no worsening or appearance of new signs and symptoms of pneumonia; there is no requirement for additional antibiotic therapy; chest roentgenograms (CT scans) are cured or improved
Time Frame: Visit 4 (within 7-9 days after last dose)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nemonoxacin | Tavanic®
Number analyzed (Participants) | 169 | 166
Participants
  Clinical success | 158 | 145
  Clinical non-efficacy | 6 | 8
  Indefinite response | 5 | 13
Statistical Analysis 1: Comparison: Nemonoxacin vs Tavanic®; Test type: Non-Inferiority — The non-inferiority bound was designated at the level of -15%; Difference in percentage = 6.1, 95% CI 2-sided [-0.7 to 13.0]
Statistical Analysis 2: Comparison: Nemonoxacin vs Tavanic®; Test type: Other; p = 0.499, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.49 to 4.29]

2. Secondary Outcome: Number of Patients With Clinical Success as Judged by the Investigator
Description: Clinical response is evaluated as clinical success if: all signs and symptoms of pneumonia are resolved or improved with no worsening or appearance of new signs and symptoms of pneumonia; there is no requirement for additional antibiotic therapy
Time Frame: Visit 2(day 4/8 ot treatment), Visit 3 (within 1-2 days after last dose)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nemonoxacin | Tavanic®
Number analyzed (Participants) | 169 | 166
Participants
  Visit 2: Clinical success | 164 | 154
  Visit 2: Clinical non-efficacy | 4 | 5
  Visit 2: Indefinite response | 1 | 7
  Visit 3: Clinical success | 160 | 151
  Visit 3: Clinical non-efficacy | 6 | 7
  Visit 3: Indefinite response | 3 | 8
Statistical Analysis 1: Comparison: Nemonoxacin vs Tavanic®; Visit 2; Test type: Other; p = 0.08, Barnard's test; Difference in percentage = 4.3, 95% CI 2-sided [-0.6 to 9.7]
Statistical Analysis 2: Comparison: Nemonoxacin vs Tavanic®; Visit 3; Test type: Other; p = 0.246, Barnard's test; Difference in percentage = 3.7, 95% CI 2-sided [-2.0 to 9.8]

3. Secondary Outcome: Number of Patients With Infection Relapse
Time Frame: Visit 5 (within 21-23 days after last dose)
Population: All patients of mITT population achieved clinical success on Visit 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nemonoxacin | Tavanic®
Number analyzed (Participants) | 158 | 145
Participants | 0 | 2
Statistical Analysis 1: Comparison: Nemonoxacin vs Tavanic®; Test type: Other; p = 0.154, Barnard test

4. Secondary Outcome: Time to Switch Therapy From Intravenous to Oral Therapy
Time Frame: Up to Visit 2 (day 4/8 ot treatment)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nemonoxacin | Tavanic®
Number analyzed (Participants) | 169 | 166
days | 4 [3 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Nemonoxacin vs Tavanic®; Test type: Other; p = 0.14, Log Rank

5. Secondary Outcome: Number of Patients Required for Other Antibiotic Treatment
Time Frame: Up to 21-23 days after last dose
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nemonoxacin | Tavanic®
Number analyzed (Participants) | 169 | 166
Participants | 2 | 5
Statistical Analysis 1: Comparison: Nemonoxacin vs Tavanic®; Test type: Other; p = 0.26, Barnard test

6. Secondary Outcome: Number of Patients With Microbiological Success
Description: Microbiological response is evaluated as microbiological success if culture study demonstrates eradication of pathogen or no material available for culture because of clinical success
Time Frame: Visit 2 (day 4/8 ot treatment), 3 (within 1-2 days after last dose), 4 (within 7-9 days after last dose)
Population: b-mITT - Patients in the mITT population whose bacterial culture had at least one baseline bacterial isolate
Measure: Count of Participants; unit: Participants
Arm/Group | Nemonoxacin | Tavanic®
Number analyzed (Participants) | 20 | 16
Participants
  Visit 2 | 17 | 16
  Visit 3 | 19 | 16
  Visit 4 | 19 | 16
Statistical Analysis 1: Comparison: Nemonoxacin vs Tavanic®; Test type: Other; p = 0.14, Barnard's test — Visit 2 assessment
Statistical Analysis 2: Comparison: Nemonoxacin vs Tavanic®; Test type: Other; p = 0.515, Barnard's test — Visit 3 assessment
Statistical Analysis 3: Comparison: Nemonoxacin vs Tavanic®; Test type: Other; p = 0.515, Barnard's test — Visit 4 assessment

7. Other Pre Specified Outcome: Nemnoxacin Concentration Changes
Description: Cmax - The peak Nemonoxacin concentration at Day 1-2 of treatment
  C-22.5hours - 22.5-h drug concentration of Nemonoxacin
Time Frame: Day 1 pre-dose and 0, 0.5, 2.5, 4, 6, 12, 16 and 22.5 (= Day 2 pre-dose) hrs after the end of first infusion on Day 1 of treatment
Population: All patients who were included in Pharmacokinetic study and who had at least 1 measured concentration value.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 15
ng/ml
  Cmax | 8163.84 (2936.57)
  C-22.5hours | 359.63 (255.88)

8. Other Pre Specified Outcome: Area Under the Concentration-time Curve (AUC) of Nemonoxacin
Description: AUC (0-22.5) - Area under the concentration-time curve from 0 to 22.5 hours of Nemonoxacin
  AUC(0-∞) - Areas under the concentration-time curve from 0 h to infinity of Nemonoxacin
Time Frame: as for outcome 7
Population: All patients who were included in Pharmacokinetic study and who had at least 1 measured concentration value.
Measure: Mean (Standard Deviation); unit: hours*ng/ml
Groups:
- Nemonoxacin: Blood sample collection for pharmacokinetic (PK) parameters was withdrawn on Day 1 and 2 of Visit 1 before and after the first infusion only in 40 first patients enrolled in the investigational sites defined by the Sponsor.
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 16
hours*ng/ml
  AUC (0-22.5) | 34372.69 (12881.56)
  AUC(0-∞) | 38560.90 (15872.29)

9. Other Pre Specified Outcome: Сlearance (CL) of Nemonoxacin
Description: Total systemic clearance of Nemonoxacin
Time Frame: as for outcome 7
Population: All patients who were included in Pharmacokinetic study and who had at least 1 measured concentration value.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 16
ml/min | 247.32 (86.92)

10. Other Pre Specified Outcome: Volume of Distribution at Steady State (Vss) of Nemonoxacin
Description: Volume of distribution at steady state of Nemonoxacin
Time Frame: as for outcome 7
Population: All patients who were included in Pharmacokinetic study and who had at least 1 measured concentration value.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 16
liters | 123.76 (39.15)

11. Other Pre Specified Outcome: Terminal Elimination Half-life (T1/2) of Nemonoxacin
Description: Terminal elimination half-life of Nemonoxacin
Time Frame: as for outcome 7
Population: All patients who were included in Pharmacokinetic study and who had at least 1 measured concentration value.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 16
hours | 7.04 (1.98)

ADVERSE EVENTS:
Time Frame: Up to 23 Days after the last dose of treatment
Arm/Group | Nemonoxacin | Tavanic®
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/169
Serious Adverse Events (participants affected / at risk) | 0/171 | 2/169
Other Adverse Events (participants affected / at risk) | 86/171 | 67/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemonoxacin (N=171) | Tavanic® (N=169)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemonoxacin (N=171) | Tavanic® (N=169)
Alanine aminotransferase increased (Investigations) | 14 (15) | 9 (9)
Platelet count increased (Investigations) | 10 (10) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 10 (10) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 6 (6)
Blood creatinine increased (Investigations) | 2 (2) | 4 (4)
Red blood cell sedimentation rate increased (Investigations) | 2 (2) | 4 (4)
Blood glucose increased (Investigations) | 3 (3) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 2 (2)
Transaminases increased (Investigations) | 3 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 6 (6)
Injection site pain (General disorders) | 4 (9) | 0 (0)
Injection site erythema (General disorders) | 3 (4) | 0 (0)
Injection site reaction (General disorders) | 3 (3) | 0 (0)
Injection site hypoaesthesia (General disorders) | 2 (4) | 0 (0)
HIV infection (Infections and infestations) | 1 (1) | 3 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT03551210/Prot_SAP_000.pdf